CLINICAL TRIAL: NCT05333419
Title: Open Label Study to Evaluate the Safety, Tolerability and Biodegradation Period of PA5346 Latanoprost Free Acid (FA) Sustained Release (SR) Ocular Implant When Administered to Patients With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Study of a Latanoprost Ocular Implant for Treatment of Open Angle Glaucoma or Ocular Hypertension.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PolyActiva Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LATA-CS103
Record Dates: First submitted 2022-03-09; First posted 2022-04-19 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Dose 100ng/day PA5346 Latanoprost FA SR Ocular Implant (Experimental): After washout, eligible subjects will be dosed with a single 100ng/day PA5346 Latanoprost FA SR Ocular Implant at study Day 0.
  Interventions: Drug: 100ng/day PA5346 Latanoprost FA SR Ocular Implant

INTERVENTIONS:
Drug: 100ng/day PA5346 Latanoprost FA SR Ocular Implant — PA5346 ocular implant is a small, clear rod-shaped implant that is placed in the anterior (front) chamber of the eye, at a single timepoint, and slowly releases a drug called latanoprost free acid (100ng/day) over a period of approximately 30 weeks

SUMMARY:
This is an open label, single dose (100 ng/day) study to assess the safety, tolerability and biodegradation of the PA5436 Latanoprost FA SR Ocular Implant in adults who have OAG or OHT.

DETAILED DESCRIPTION:
Participants who are currently administering Intraocular Pressure lowering drop therapy for Open Angle Glaucoma or Ocular Hypertension will be recruited.

Prior to recruitment, participants will be medicated with IOP lowering drop therapy, including a prostaglandin analogue to manage their POAG. The IOP lowering eye drops will be stopped in the intent to treat (ITT) eye at least 28 days and no greater than 49 days prior to the date of implant administration.

Participants will be required to have an unmedicated (post washout) 8:00 AM IOP ≥ 24 mmHg and ≤ 36 mmHg in the ITT eye at either of 2 screening visits 2 weeks apart.

Participants are also required to have an unmedicated (post washout) IOP ≥ 20 mmHg and ≤ 36 mmHg at 12:00 noon and 4:00 PM in the same eye on the same screening visit where the 8:00 AM IOP was IOP ≥ 24 mmHg and ≤ 36mmHg.

The PA5346 Latanoprost FA SR Ocular Implant will be administered to one eye (unilateral) of each participant.

IOP will be monitored and if during the course of the study it is found to rise ≥ 30% over baseline in the study eye(s), IOP lowering eye drops will be resumed.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
* Diagnosis of OAG or OHT. Iridocorneal angle must be classified as Grade 3 or 4 on the modified Shaffer-Etienne scale by gonioscopy.
* Unmedicated (post-washout) 8:00 AM IOP of 24 mmHg to 36 mmHg in the ITT eye at either of two qualification visits 2 weeks apart. In addition, the IOP at 12:00 noon and 4:00 PM must be 20 mmHg to 36 mmHg on the same qualification visit where the 8:00 AM IOP was IOP 24 mmHg to 36 mmHg.
* Have a corrected visual acuity as determined by Early Treatment of Diabetic Retinopathy Study (ETDRS) charts in each eye greater than or equal to + 0.3 logMAR (equivalent to 6/12).
* Minimum central endothelial cell density of greater than or equal to 1600 cells/mm2 as determined by the reading centre adopted for the study.
* Currently managing their OAG or OHT with IOP lowering drop therapy, including a prostaglandin analogue.
* Are able and willing to follow study instructions and adhere to the protocol schedule and restrictions and undergo eye examinations

Exclusion Criteria:

* Have pseudoexfoliation or pigment dispersion glaucoma
* Have aphakic eyes or only one functioning eye. only one eye.
* Have had iIntraocular surgery, glaucoma surgery or cornea/refractive surgery within the past 6 months or anticipate a need for eye surgery (including laser) in the study eye during the study period. .
* Significant corneal guttatae
* Ocular trauma in either eye within the three months prior to screening
* Current retinal detachment or history of blunt trauma in the study eye.
* Clinically significant ocular disease in either eye (e.g., corneal oedema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study Ocular trauma
* Have a known sensitivity to any component of the product (e.g. latanoprost, or polytriazole sensitivity), or to topical therapy used during the course of the study. Ocular infection or inflammation
* Have a clinical diagnosis of Fuchs' Endothelial Corneal Dystrophy (FECD) in the study eye or have confluent central corneal guttatae, multiple central guttatae greater than a single cell, or corneal disease or abnormality that would prevent specular microscopy corneal scans of the study eye.
* Central corneal thickness in either eye that is less than 470 µm or greater than 630 µm at screening (or a difference between the eyes >70 µm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of 100 ng/day PA5346 Latanoprost FA SR Ocular Implant in adults with Open Angle Glaucoma (OAG) or Ocular Hypertension (OHT). | Change from baseline to 40 weeks
  Clinically significant changes to haematology or biochemistry
To assess the safety and tolerability of 100 ng/day PA5346 Latanoprost FA SR Ocular Implant in adults with Open Angle Glaucoma (OAG) or Ocular Hypertension (OHT). | Change from baseline to 40 weeks
  Clinically significant changes to urinalysis
To assess the safety and tolerability of 100 ng/day PA5346 Latanoprost FA SR Ocular Implant in adults with Open Angle Glaucoma (OAG) or Ocular Hypertension (OHT). | Change from baseline to 40 weeks
  Clinically significant changes to physical examination
To assess the safety and tolerability of 100 ng/day PA5346 Latanoprost FA SR Ocular Implant in adults with Open Angle Glaucoma (OAG) or Ocular Hypertension (OHT). | Change from baseline to 40 weeks
  Clinically significant changes to vital signs
To assess the safety and tolerability of 100 ng/day PA5346 Latanoprost FA SR Ocular Implant in adults with Open Angle Glaucoma (OAG) or Ocular Hypertension (OHT). | Change from baseline to 40 weekls
  Clinically significant changes to visual acuity
To assess the period of biodegradation of 100 ng/day PA5346 Latanoprost FA SR Ocular Implant in adults with OAG or OHT. | Up to 12 months
  Biodegradation will be assessed by Gonioscopy or anterior Optical Coherence at Tomography (OCT) at Weeks 6, 12, 18, 26, 34, 40 and each subsequent 6 week visit thereafter until the implant has completely biodegraded. These tests allow the implant to be located by the ophthalmologist.

SECONDARY OUTCOMES:
To assess the initial efficacy of 100 ng/day PA5346 Latanoprost FA SR Ocular Implant in controlling IOP during a study period in adults with OAG or OHT. | Up to 12 months
  IOP will be assess by using a tonometer at Day 1, Weeks 6, 18, 26, 34, 40 and every 6 weekly visit after intervention commencement.
Extent of hyperaemia. | Up to 12 months
  Assessed by Slit lamp Biomicroscopy for Conjunctival Redness Day 1, Weeks 6, 18, 26, 34, 40 and every 6 weekly visit after intervention commencement.
Ophthalmologist-reported ease of use of bespoke administration device | Day 0
  This questionnaire is descriptive only and includes questions such as:
  * Ease of attaching the implant-containing needle to the administration device
  * Ease of inserting the implant in the correct location
  * Number of times the plunger is depressed to extrude the implant.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Wells, MD, Principal Investigator — Capital Eye Specialists
Locations (2):
- New Zealand (2):
  - Capital Eye Specialists, Te Aro, Wellington Region
  - Rotorua Eye Clinic, Rotorua

IPD SHARING:
Plan to Share IPD: No